CLINICAL TRIAL: NCT00494039
Title: I-125 Versus Pd-103 for Low Risk Prostate Cancer
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: VA Puget Sound Health Care System (U.S. Federal Agency)
Collaborators: Schiffler Cancer Center (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IP
Record Dates: First submitted 2007-06-28; First posted 2007-06-29 (Estimated); Last update posted 2007-06-29 (Estimated); Status verified 2007-06

CONDITIONS: Prostate Cancer
Keywords: prostate; cancer; radiation; brachytherapy
MeSH Terms: conditions — Prostatic Neoplasms; Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Procedure: Radioactive seed implant to prostate

SUMMARY:
Objective: To test the hypothesis that the shorter half-life of Pd-103 versus I-125, will increase the rate of tumor eradication.

Research design A total of 600 patients with AJC clinical stage T1c-T2a prostatic carcinoma (Gleason grade 2 to 6, PSA 4 to 10 ng/ml) will be randomized to implantation with I-125 (160 Gy) versus Pd-103 (115 Gy).

DETAILED DESCRIPTION:
Objective: To test the hypothesis that the shorter half-life of Pd-103 versus I-125, will increase the rate of tumor eradication.

Research design A total of 600 patients with AJC clinical stage T1c-T2a prostatic carcinoma (Gleason grade 2 to 6, PSA 4 to 10 ng/ml) will be randomized to implantation with I-125 (160 Gy) versus Pd-103 (115 Gy).

Methodology: Patients will be randomized by the method of random permuted blocks.

Cancer status will be monitored by serial serum PSA at 6, 12, 18 and 24 months and yearly thereafter. Treatment-related morbidity will be monitored by personal interview, using standard American Urologic Association and Radiation Therapy Oncology Group criteria at 1, 3, 6, 12 and 24 months. Patients with serum PSA above 1.0 ng/ml two years after treatment will be considered to have residual or recurrent cancer and to have failed therapy.

ELIGIBILITY:
Inclusion Criteria:

* Males age 40-80
* PSA 4-10
* Gleason score 5-6

Exclusion Criteria:

* Lymph node positive

Ages: 40 Years to 80 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 602 (Actual)
Dates: Start 1998-01; Study Completion 2010-01 (Estimated)

PRIMARY OUTCOMES:
Cancer control (biochemical and survival) | final analysis 2008(?)

CONTACTS AND LOCATIONS:
Overall Officials: Kent E Wallner, MD, Study Chair — Puget Sound Health Care system
Locations (1):
- Puget Sound VA, Seattle, Washington, United States

REFERENCES:
- [Result] Wallner K, Merrick G, True L, Sutlief S, Cavanagh W, Butler W. 125I versus 103Pd for low-risk prostate cancer: preliminary PSA outcomes from a prospective randomized multicenter trial. Int J Radiat Oncol Biol Phys. 2003 Dec 1;57(5):1297-303. doi: 10.1016/s0360-3016(03)01448-2. PMID 14630265
- [Result] Wallner K, Merrick G, True L, Cavanagh W, Simpson C, Butler W. I-125 versus Pd-103 for low-risk prostate cancer: morbidity outcomes from a prospective randomized multicenter trial. Cancer J. 2002 Jan-Feb;8(1):67-73. doi: 10.1097/00130404-200201000-00012. PMID 11895205